CLINICAL TRIAL: NCT02180412
Title: A Double-blind, Randomized, Placebo-controlled, Parallel Group Trial on the Efficacy and Safety of PanhematinTM in the Treatment of Acute Attacks of Porphyria
Brief Title: Controlled Trial of Panhematin in Treatment of Acute Attacks of Porphyria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10-203; FD-R-03720 (Other Grant/Funding Number: FDA OOPD)
Record Dates: First submitted 2014-06-25; First posted 2014-07-02 (Estimated); Results first posted 2025-04-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Porphyrias
Keywords: Acute porphyria; Hemin
MeSH Terms: conditions — Porphyria, Acute Intermittent | interventions — Hemin; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Panhematin (Experimental): Panhematin plus glucose
  Interventions: Biological: Panhematin; Other: Glucose
- Placebo (Placebo Comparator): Placebo (saline) plus glucose
  Interventions: Other: Glucose

INTERVENTIONS:
Biological: Panhematin — Glucose loading
  Other Names: Glucose
  Arms: Panhematin
Other: Glucose — Glucose is administered to both groups as routine care.

SUMMARY:
This study aims to provide high quality evidence for the effectiveness and safety of hemin (PanhematinTM , Recordati) for treatment of acute attacks of porphyria. These types of studies have not been done before with either PanhematinTM or the hemin preparation available in Europe (NormosangTM, Orphan Europe).

There are two treatment groups in this study. One group will be treated with PanhematinTM plus glucose, and the other group will be treated with glucose plus an inactive salt solution (called a "placebo"). To avoid prejudice, the treatment given to each participant will be blinded (meaning the participants and most of the hospital staff will not know which treatment the participant will receive) and randomized (meaning participants will have an equal chance of receiving either treatment, like the flip of a coin). A placebo-controlled, randomized study is the standard method used to prove treatments are effective and safe. PanhematinTM and glucose will be given in the same manner as is usual for treating an attack of porphyria. For participants who are chosen to receive the placebo, their treatment will be switched to real PanhematinTM at any time if their symptoms do not improve. This is called "rescue" treatment, and assures that they study is safe and patients who need hemin will receive it. Treatment with hemin will be for 4 days, or longer if needed. Since the study treatment is started as soon as possible after symptoms appear, there will be very little delay in providing hemin to those who need it. Funding Source - Office of Orphan Products Development (FDA OOPD)

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 years
* Willing to provide written informed consent
* Acute symptoms (7 days duration or less to time of enrollment) such as abdominal, back and/or limb pain, diagnosed by the investigator as caused by porphyria after initial evaluation has excluded other causes.
* Diagnosis of acute porphyria documented by a substantial increase in urinary or serum porphobilinogen (PBG).
* Type of acute porphyria confirmed by additional testing (in addition to increased PBG), which may be completed before or after treatment begins using pretreatment samples:
* For acute intermittent porphyria (AIP): Normal or only slight increases in plasma and fecal porphyrins. Most (~90 percent) will have deficient activity of erythrocyte porphobilinogen deaminase (PBGD), and almost all (>95 percent) will have a demonstrable disease-causing PBGD mutation.
* For hereditary coproporphyria (HCP): Substantial increases in fecal porphyrins (almost entirely coproporphyrin III). In the absence of skin photosensitivity, most will have normal or only slight increases in plasma porphyrins. Almost all (>95 percent) will have a demonstrable disease-causing coproporphyrinogen oxidase (CPO) mutation.
* For variegate porphyria (VP): Substantial increases in fecal porphyrins (mostly coproporphyrin III and protoporphyrin), increased plasma total porphyrins and a fluorescence emission maximum of diluted plasma at neutral pH near 626 nm. Almost all (~95 percent) will have a demonstrable disease-causing protoporphyrinogen oxidase (PPO) mutation.

Exclusion Criteria:

* Symptoms such as abdominal, back or limb pain are explained by another condition, as judged by the investigator
* Therapy with hemin within 7 days prior to enrollment in this study
* Known or suspected allergy to Panhematin™ or related products
* Preexisting coagulation defect or concurrent treatment with an anticoagulant
* Previously documented renal impairment defined as a serum creatinine above 1.7 mg/dL or 150 mmol/L.
* A diagnosis of diabetes mellitus, which might increase the risk of glucose infusion.
* Heart failure, significant chronic anemia or any disease or condition that the investigator judges would lead to an unacceptable risk to the patient or interfere with the successful collection of date for the trial
* Previous randomization in this trial

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-04-28 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karl E Anderson, MD, Principal Investigator — UT, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Panhematin | Placebo
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Panhematin | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.6 (6.2) | 36.7 (11.2) | 36.7 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 20
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 0 | 1 | 1
  Non-Hispanic American Indian or Alaskan native | 1 | 0 | 1
  Non-Hispanic Asian | 0 | 1 | 1
  Non-Hispanic Black or African American | 0 | 2 | 2
  Non-Hispanic White | 9 | 6 | 15

OUTCOME MEASURES:

1. Primary Outcome: Difference in NRS Pain Score Between Baseline and 12 Hours
Description: The difference in the pre-infusion NRS pain scores and NRS pain score 12 hours from the infusion start time. To define this variable, all blinded study treatment infusion times were compared with the pain score survey times. The pain score closest to but prior to the infusion time was the pre-infusion pain score. Numeric rating scale for pain (0-10; 0=no pain, 10=most severe pain).
Time Frame: Baseline and 12 hours
Population: One participant was randomized incorrectly and didn't meet inclusion criteria. Therefore, this analysis was done without one participant, making this analysis done under modified intent-to-treat protocol, not true intent-to-treat protocol.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Panhematin | Placebo
Number analyzed (Participants) | 9 | 10
score on a scale | -0.2 (2.2) | -0.2 (1.9)

2. Secondary Outcome: Biochemical Effects of Panhematin In Participants Treated Early For Attacks of Porphyria
Description: Difference in the panhematin and placebo arm for the change in urinary ALA, (PBG), and total porphyrins between baseline and subsequent time points.
Time Frame: Day 1 (baseline), Day 2, Day 3 and Day 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mean difference of mg/g creatinine
Arm/Group | Panhematin | Placebo
Number analyzed (Participants) | 9 | 10
mean difference of mg/g creatinine
  ALA Day 1 vs Day 2 | 8.47 (8.97) | 2.31 (5.5)
  ALA Day 1 vs Day 3 | 13.27 (11.45) | -0.57 (6.01)
  ALA Day 1 vs Day 4 | 14.90 (11.85) | 1.99 (10.73)
  PBG Day 1 vs Day 2 | 6.56 (11.69) | -2.94 (12.85)
  PBG Day 1 vs Day 3 | 15.56 (17.88) | -7.08 (10.76)
  PBG Day 1 vs Day 4 | 20.16 (18.63) | -5.83 (20.00)
  Total Porphyrins Day 1 vs Day 2 | 297.60 (948.90) | 317.00 (682.93)
  Total Porphyrins Day 1 vs Day 3 | 594.00 (1173.48) | 165.00 (678.41)
  Total Porphyrins Day 1 vs Day 4 | 606.11 (1238.87) | 331.33 (836.59)
Statistical Analysis 1: Comparison: Panhematin vs Placebo; ALA Day 1 vs Day 2; Test type: Other; p = .0434, ANCOVA; Slope = 7.76, 95% CI 2-sided [2.14 to 13.37]
Statistical Analysis 2: Comparison: Panhematin vs Placebo; ALA Day 1 vs Day 3; Test type: Other; p = .0003, ANCOVA; Slope = 16.29, 95% CI 2-sided [11.32 to 21.25]
Statistical Analysis 3: Comparison: Panhematin vs Placebo; ALA Day 1 vs Day 4; Test type: Other; p = .0198, ANCOVA; Slope = 15.98, 95% CI 2-sided [6.7 to 25.26]
Statistical Analysis 4: Comparison: Panhematin vs Placebo; PBG Day 1 vs Day 2; Test type: Other; p = .158, ANCOVA; Slope = 10.69, 95% CI 2-sided [-1.67 to 22.49]
Statistical Analysis 5: Comparison: Panhematin vs Placebo; PGB Day 1 vs Day 3; Test type: Other; p = .0127, ANCOVA; Slope = 24.52, 95% CI 2-sided [11.3 to 37.74]
Statistical Analysis 6: Comparison: Panhematin vs Placebo; PBG Day 1 vs Day 4; Test type: Other; p = .0328, ANCOVA; Slope = 28.45, 95% CI 2-sided [9.64 to 47.27]
Statistical Analysis 7: Comparison: Panhematin vs Placebo; Total Porphyrins Day 1 vs Day 2; Test type: Other; p = .9993, ANCOVA; Slope = 12.2, 95% CI 2-sided [-465.4 to 489.8]
Statistical Analysis 8: Comparison: Panhematin vs Placebo; Total Porphyrins Day 1 vs Day 3; Test type: Other; p = .2915, ANCOVA; Slope = 454.5, 95% CI 2-sided [-200.87 to 1109.86]
Statistical Analysis 9: Comparison: Panhematin vs Placebo; Total Porphyrins Day 1 vs Day 4; Test type: Other; p = .4382, ANCOVA; Slope = 326.12, 95% CI 2-sided [-292 to 944.25]

3. Other Pre Specified Outcome: Effects of Clinical Features on Response to Panhematin
Description: Age, sex, exacerbating factors
Time Frame: 4 days
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Effects of Genetic Features on Response to Panhematin
Description: Types of mutations
Time Frame: 4 days
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Use of Reconstitution of Panhematin With Albumin
Description: Frequency of side effects or adverse events
Time Frame: 4 days
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 1 (baseline), Day 2, Day 3 and Day 4
Arm/Group | Panhematin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 0/10 | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-02): https://cdn.clinicaltrials.gov/large-docs/12/NCT02180412/Prot_SAP_000.pdf